CLINICAL TRIAL: NCT03843775
Title: A Phase I/II Study of Binimetinib With Encorafenib in Patients With Non-V600 Activating BRAF Mutant Advanced Malignancies
Brief Title: A Study of Binimetinib and Encorafenib in Advanced BRAF Mutant Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-547
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Advanced BRAF Mutant Cancers
Keywords: Binimetinib; Encorafenib; 18-547
MeSH Terms: interventions — binimetinib; encorafenib

STUDY DESIGN:
Intervention Model Description: This phase I/II study consists of a Phase I part followed by an efficacy analysis (Phase II) of the dosing schedule deemed safe in patients with advanced cancer with activating non-V600 BRAF mutant tumors. As patients in the phase I part of the start will start at the lower dose level 1, they will not be included in the stage one efficacy cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Binimetinib and Encorafenib (Experimental): Patients will be initially enrolled to the approved dose of encorafenib 450 mg oral QD and binimetinib 45 mg PO BID, dose level 1. If confirmed this dose level is safely tolerated in the study population, we will then escalate treatment to dose level 2 with the novel dosing regimen of encorafenib 450 mg oral QD continuous and binimetinib 60 mg oral BID 21 days on/7 days off.
  Interventions: Drug: Binimetinib; Drug: Encorafenib

INTERVENTIONS:
Drug: Binimetinib — Dose level 1 binimetinib 45 mg PO BID. Dose level 2 binimetinib 60 mg oral BID
  Other Names: MEK162 or ARRY-438162
Drug: Encorafenib — encorafenib 450 mg oral QD
  Other Names: LGX818

SUMMARY:
The goal of this trial is to test the safety and efficacy of an innovative combination aimed to more profoundly inhibit ERK signaling in tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed the Informed Consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements
* Age ≥ 18 years at the time of informed consent
* Metastatic or advanced-stage malignant tumors confirmed histologically for whom no standard therapy is considered to be appropriate by the investigator
* Patients must have at least one other lesion that is measurable by RECIST criteria.
* Patient's tumor must harbor an activating BRAF mutation (listed in Table 4 or approved by the study Principal Investigator) or a fusion involving the kinase domain of BRAF
* Mechanistically validated activating non-V600 BRAF mutants

  * P367L/S
  * G464V/E
  * G469A/V/R
  * L485W
  * N486_A489delinsK
  * N486_P490del
  * E586K
  * L597Q/V/S
  * T599TT/TS
  * T599I/K
  * V600_K601delinsE
  * K601E/N/T
  * K601_S602delinsNT
  * BRAF kinase duplication
  * Fusions involving BRAF kinase domain
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Adequate bone marrow, organ function and laboratory parameters:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Hemoglobin (Hgb) ≥ 8 g/dL with or without transfusions
  * Platelets (PLT) ≥ 75 x 109/L without transfusions
  * AST and/or ALT ≤ 2.5 × upper limit of normal (ULN); patient with liver metastases ≤ 5 ×ULN
  * Total bilirubin ≤ 1.5 × ULN and < 2 mg/dL (Note: Patients who have a total bilirubin level > 1.5 x ULN will be allowed if their indirect bilirubin level is ≤ 1.5 x ULN)
  * Serum Creatinine ≤ 1.5 x ULN, or calculated creatinine clearance (determined as per Cockcroft-Gault) ≥ 50 mL/min at screening
* Adequate cardiac function:

  * left ventricular ejection fraction (LVEF) ≥ 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram
  * QTc interval ≤ 480 ms (preferably the mean from triplicate ECGs)
* Able to take oral medications
* Patient is deemed by the Investigator to have the initiative and means to be compliant with the protocol (treatment and follow-up)
* Female patients are either postmenopausal for at least 1 year, are surgically sterile for at least 6 weeks, or must agree to take appropriate precautions to avoid pregnancy from screening through 30 days after the last dose of study drug/treatmentif of childbearing potential (Note: Permitted contraception methods listed in Section 9.3 should be communicated to the patients and their understanding confirmed. For females of childbearing potential, the pregnancy test result must be negative at screening.)
* Males must agree to take appropriate precautions to avoid fathering a child from screening through 90 days following the end of therapy. (Note: Permitted contraception methods listed in Section 9.3 should be communicated to the patients and their understanding confirmed.)

Exclusion Criteria:

* Any symptomatic brain metastasis (Note: Patients previously treated or untreated for this condition who are asymptomatic in the absence of corticosteroid and antiepileptic therapy are allowed. Brain metastases must be stable for ≥ 4 weeks, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT]) demonstrating no current evidence of progressive brain metastases at screening.)
* History or current evidence of retinal vein occlusion (RVO) or current risk factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease
* Leptomeningeal disease
* Previous or concurrent malignancy within 2 years of study entry, with the following exceptions: adequately treated basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, early stage breast cancer, or other noninvasive or indolent malignancy
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) < 6 months prior to screening
  * Symptomatic chronic heart failure (i.e. Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia
* Uncontrolled hypertension defined as persistent elevation of systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg, despite current therapy.
* Known positive serology for HIV (Human Immunodeficiency Virus), active hepatitis B, and/or active hepatitis C infection
* Impaired GI function or disease that may significantly alter the absorption of encorafenib or binimetinib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption)
* History of thromboembolic or cerebrovascular events ≤ 12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli.

Note: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks. Note: Patients with thromboembolic events related to indwelling catheters or other procedures may be enrolled.Concurrent neuromuscular disorder that is associated with the potential of elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).

* Any other condition that would, in the Investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medications, social/psychological issues, etc.
* Patients who have undergone surgery ≤ 3 weeks prior to starting study drug or who have not yet recovered from side effects of such procedure
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Medical, psychiatric, cognitive, or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
* Prior treatment with any RAF, MEK, or ERK inhibitors (such as vemurafenib, dabrafenib, encorafenib; trametinib, cobimetinib, binimetinib, selumetinib; or BVD-523, respectively)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rona Yaegar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- [Derived] Rajkumar S, Berry D, Heney KA, Strong C, Ramsay L, Lajoie M, Alkallas R, Nguyen TT, Thomson C, Ahanfeshar-Adams M, Dankner M, Petrella T, Rose AAN, Siegel PM, Watson IR. Melanomas with concurrent BRAF non-p.V600 and NF1 loss-of-function mutations are targetable by BRAF/MEK inhibitor combination therapy. Cell Rep. 2022 Apr 5;39(1):110634. doi: 10.1016/j.celrep.2022.110634. PMID 35385748
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Encorafenib 450 mg oral QD and Binimetinib 45 mg PO BID
- Dose Level 2: Encorafenib 450 mg oral QD and Binimetinib 60 mg oral BID
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 4 | 13
Completed | 1 | 5
Not Completed | 3 | 8
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 2 | 6
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 4 | 13 | 17
Age, Continuous [Median (Full Range); unit: years] | 66 [55 to 71] | 65 [36 to 80] | 65 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 2 | 7 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 11 | 14
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 11 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 13 | 17

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities (DLTs)
Description: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 5,
Time Frame: 1 year
Population: DLTs only evaluated for Dose Level 1 cohort
Measure: Number; unit: DLTs
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 4 | 0
DLTs | 0 |

2. Primary Outcome: Objective Response Rate (Phase II)
Description: Per RECIST Version 1.1
Time Frame: 1 year
Population: ORR was only assessed for the Dose Level 2 group
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 13
percentage of participants |  | 6.7 [0.3 to 31.9]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Level 1 | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 4/4 | 12/13
Serious Adverse Events (participants affected / at risk) | 1/4 | 3/13
Other Adverse Events (participants affected / at risk) | 4/4 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=13)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=13)
Nausea (Gastrointestinal disorders) | 1 | 7
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 2
Blurred vision (Eye disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 4
Dry eye (Eye disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Thrombotic event (Vascular disorders) | 1 | 0
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 6
Alkaline phosphatase increased (Investigations) | 0 | 5
Creatinine phosphokinase increased (Investigations) | 0 | 4
Subretinal fluid (Eye disorders) | 0 | 4
AST increase (Investigations) | 0 | 4
ALT increase (Investigations) | 0 | 4
Creatinine kinase (Investigations) | 0 | 3
Fatigue (General disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Central serous chorioretinopathy (Eye disorders) | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous nodules (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Impetigo (Skin and subcutaneous tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03843775/Prot_SAP_000.pdf